CLINICAL TRIAL: NCT05704920
Title: A Randomized Controlled Study of Including a Deep Learning-based Analysis of Chest Computed Tomography as an Aid to Decision Making of Multidisciplinary Team Meetings for Lung Cancer Screening in Eligible Patients
Brief Title: Integrating Artificial Intelligence Into Lung Cancer Screening.
Acronym: DACAPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-PP-12
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IA Group (Experimental): Patients with at least one nodule (> 6mm) for whom the multidisciplinary team meeting discussion is informed of the AI-based analysis of their chest computed tomography
  Interventions: Other: IA
- Group not IA analysis (Other): Patients with at least one nodule (> 6mm) for whom the multidisciplinary team meeting discussion is not informed of the AI-based analysis of their chest computed tomography
  Interventions: Other: Not IA

INTERVENTIONS:
Other: IA — The multidisciplinary team meeting discussion is informed of the AI-based analysis of their chest computed tomography
  Arms: IA Group
Other: Not IA — The multidisciplinary team meeting discussion is not informed of the AI-based analysis of their chest computed tomography
  Arms: Group not IA analysis

SUMMARY:
Lung cancer (LC) screening using low-dose chest CT (LDCT) has already proven its efficacy.

The mortality reduction associated with LC screening is around 20%, much higher than the reduction in mortality associated with screening for breast, colon or prostate cancers.

Implementing lung cancer screening on a large scale faces two main obstacles:

1. The lack of thoracic radiologists and LDCT necessary for the eligible population (between 1.6 and 2.2 million people in France);
2. The high frequency of false positive screenings: in the NLST trial, more than 20% of the subjects screened were found to have at least one nodule of an indeterminate lung nodule (ILN) whereas less than 3% of ILNs are actually LC.

The gold standard for determining on the benign or malignant nature of a nodule is definitive histology. Otherwise, the evolution of the nodule on serial thoracic imaging is a good alternative. The period of indeterminacy of a nodule can be as long as 24 months in many cases, which can be a source of prolonged and sometimes unjustified anxiety for screening candidates.

The purpose of this randomized controlled study that focuses on LC screening in patients aged 50 to 80 years, who smoked more than 20 packs/ year or stopped smoking less than 15 years ago. Its objective is to determine whether assisting multidisciplinary team (MDT) meetings with an AI-based analysis of screening LDCT accelerates the definitive classification of nodules into malignant or benign.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 80 years old
* active smoker or ex-smoker who quit smoking less than 15 years ago
* smoking history of at least 20 pack-years
* signature of the informed consent
* affiliation to French social security

Exclusion Criteria:

* clinical signs suggestive of cancer
* recent chest scan (<1 year) for another cause
* radiological abnormality requiring follow-up or additional investigations
* health problem significantly limiting life expectancy from the clinician's point of view
* health problem limiting ability or willingness to undergo lung surgery
* Patients with active neoplasia, except basal cell carcinoma of the skin.
* vulnerable people: adults under guardianship, adults under curatorship medical and/or psychiatric problems of sufficient severity to limit full adherence to the study or expose patients to excessive risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2722 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of lung disease | At 3 years
  Elapsed time between lung nodule discovery and MDT decision making.

SECONDARY OUTCOMES:
Operating characteristics of Ai-based strategy | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marquette Charles-Hugo, Principal Investigator — CHU de Nice, Service de Pneumologie
Locations (1):
- CHU de Nice - Hôpital de Pasteur, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request

REFERENCES:
- [Derived] Benzaquen J, Hofman P, Lopez S, Leroy S, Rouis N, Padovani B, Fontas E, Marquette CH, Boutros J; Da Capo Study Group. Integrating artificial intelligence into lung cancer screening: a randomised controlled trial protocol. BMJ Open. 2024 Feb 13;14(2):e074680. doi: 10.1136/bmjopen-2023-074680. PMID 38355174